CLINICAL TRIAL: NCT03625830
Title: A Randomized, Multicenter Study on the Efficacy and Safety of Paclitaxel-eluting PTCA-Balloon Catheter(SeQuent® Please) Compared to POBA in the Treatment of Small Vessel Disease (SVD) Patient
Brief Title: The Efficacy and Safety of SeQuent® Please in the Treatment of Small Vessel Disease (SVD) Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-1518
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-08

CONDITIONS: Small Vessel Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel-eluting PTCA-Balloon Catheter(SeQuent® Please) (Experimental)
  Interventions: Device: Paclitaxel-eluting PTCA-Balloon Catheter(SeQuent® Please)
- Rapid exchange PTCA Balloon Catheter (SeQuent® Neo) (Active Comparator)
  Interventions: Device: rapid exchange PTCA -Balloon Catheter (SeQuent® Neo)

INTERVENTIONS:
Device: Paclitaxel-eluting PTCA-Balloon Catheter(SeQuent® Please) — SeQuent® Please in length of 10 mm, 15 mm, 17 mm, 20 mm, 26 mm, 30 mm and in diameter of 2.0 mm, 2.5mm, 2.75mm will be used in the trial.
  Arms: Paclitaxel-eluting PTCA-Balloon Catheter(SeQuent® Please)
Device: rapid exchange PTCA -Balloon Catheter (SeQuent® Neo) — SeQuent® Please in length of 10 mm, 15 mm, 17 mm, 20 mm, 26 mm, 30 mm and in diameter of 2.0 mm, 2.5mm, 2.75mm will be used in the trial.
  Arms: Rapid exchange PTCA Balloon Catheter (SeQuent® Neo)

SUMMARY:
The purpose is to evaluate the safety and effectiveness of paclitaxel-releasing coronary balloon (Catheter SeQuent® Please) versus rapid exchange PTCA balloon catheter (SeQuent® Neo) in the treatment of stenoses of coronary small vessels. 270 subjects will be enrolled for the trials.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to subjects

* Patients with stable angina pectoris, or unstable angina pectoris, or old myocardial infarction, or documented silent ischemia;
* At the age of 18-80;
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the study. Hence, patients will be advised to use an adequate birth control method up to (including) the end of follow-up;
* Patients must agree to undergo the 9-month angiographic follow-up and the clinical follow-up at 30 days, 6 months, 9 months and 12 months after operation;
* Patients who are psychologically and linguistically able to understand the purpose of the study, and show sufficient compliance with the study protocol;
* Patients who have expressed acknowledgment of the risks and benefits described in the informed consent document by providing informed consent;

Criteria related to lesions

* The target lesion is primary, in situ coronary artery lesion located in 1 or 2 different coronary arteries, with no more than 1 target lesion in each coronary artery;
* The reference vessel diameter is within the range of 2.0 mm - 2.75 mm; (visually measured)
* Interventional treatment should be conducted on lesion(s) of non-target vessel(s) in advance (which must be concurrent treatment), and management of random and target lesions should be performed after successful treatment of non-target lesion(s);
* The pre-operative diameter stenosis must be either ≥ 70% or ≥ 50% with ischemia; (visually measured)
* Each target lesion should be treated with only one SeQuent® Please or SeQuent® Neo.

Exclusion Criteria:

Criteria related to subjects

* Patients with recent myocardial infarction (within one week), or patients with myocardial infarction over one week but whose troponin level has not recovered to normal;
* Patients with severe congestive heart failure or NYHA class IV heart failure;
* Patients with severe valvular heart disease;
* Women who are pregnant or lactating;
* Patients with remaining life expectancy of no more than 1 year or with factors causing difficulty in clinical follow-up;
* Patients who had cerebral stroke within 6 months before operation;
* Patients who are currently involved in any other clinical trial;
* Patients with presence or history of severe hepatic failure and therefore are not eligible for angiography;
* Patients with presence or history of severe renal failure (GFR < 30 ml/min) and therefore are not eligible for angiography;
* Patients who have received heart transplant;
* Patients with cardiogenic shock;
* Patients with left ventricular ejection fraction less than 30%;
* Patients suffering from coronary artery spasm without significant stenosis;
* Patients considered as ineligible by the investigator for other reasons;

Criteria related to lesions

* Evidence of extensive thrombosis in target vessel before intervention;
* Percutaneous coronary intervention of venous graft;
* Chronic total occlusion (TIMI 0 flow before operation);
* Left main disease and/or triple vessel disease needed to be treated, bifurcation lesion with branch vessel diameter ≥ 2.5 mm, and bypass graft lesion;
* There is non-target lesion(s) in the proximal large vessel and target lesion(s) in the distal small vessel of the same vessel (eligible if there is non-target lesion(s) in proximal large vessel and a target lesion in the bifurcated small vessel);
* The target vessel is distorted or has calcified lesion(s);
* Lesion within 5 mm away from the coronary artery ostium;
* Lesion that cannot be treated with PTCA or other interventional techniques;
* After pre-dilation of target lesion, the residual stenosis is ≥ 30% or TIMI flow is < 3, and/or type C or above dissection appears;

Exclusion criteria related to concomitant medication

* Patients prone to bleeding and contraindicated for anticoagulant or antiplatelet drugs;
* Patients who are intolerant to aspirin and/or clopidogrel or have a history of neutrophilopenia or thrombocytopenia, or patients with severe hepatic insufficiency and contraindicated for clopidogrel.
* Patients who are known to be intolerant or allergic to heparin, contrast agent, paclitaxel, iopromide, rapamycin, polylactic acid - glycolic acid polymer, stainless steel;
* Patients with a history of leukopenia (leukocyte count < 3 × 109/L for more than 3 days), neutrophilopenia (ANC < 1,000 neutrophils/mm3 for more than 3 days), or thrombocytopenia (< 100,000 platelets/mm3);
* Patients with a history of peptic ulcer or gastrointestinal bleeding in the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss in segment section at M9 | 9 months
  To measure the diameter loss in the in-segment late lumen loss (LLL) at 9 months after operation by using angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu K, Fu X, Yang W, Wu Y, Li C, Ding D, Wang Z, Chu M, Qian J, He B, Tu S, Shen L, Ge J. A novel angiographic index for predicting the efficacy of drug-coated balloons in small vessels. EuroIntervention. 2025 Oct 20;21(20):e1209-e1221. doi: 10.4244/EIJ-D-25-00075. PMID 41117656